CLINICAL TRIAL: NCT02648932
Title: The Rapid Study: Randomized (RA) Phase (P) II Study To Expedite Allogeneic Transplant With Immediate (I) Haploidentical Plus Unrelated Cord Donor (D) Search Versus Matched Unrelated Donor Search For AML And High-Risk MDS Patients
Brief Title: The Rapid Study: Randomized Phase II Study To Expedite Allogeneic Transplant With Immediate Haploidentical Plus Unrelated Cord Donor Search Versus Matched Unrelated Donor Search For AML And High-Risk MDS Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB15-0866
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-02

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
Keywords: Acute Myeloid Leukemia (AML); High-Risk Myelodysplastic Syndrome (MDS); hematopoietic cell transplantation; haplo-cord search; matched unrelated donor search
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haplo-Cord Search (Other): If subject meets the inclusion criteria and consents, will undergo a haplo-cord transplant.
  Interventions: Biological: Haplo-Cord Transplant
- Matched Unrelated Donor Search (MUD) (Other): If subject meets the inclusion criteria and consents, will undergo a MUD transplant.
  Interventions: Procedure: Matched Unrelated Donor Transplant

INTERVENTIONS:
Biological: Haplo-Cord Transplant — For conditioning regimens, haplo-identical grafts will be selected by the Miltenyi Device
  Arms: Haplo-Cord Search
Procedure: Matched Unrelated Donor Transplant
  Arms: Matched Unrelated Donor Search (MUD)

SUMMARY:
The study seeks to compare time from formal search to hematopoietic cell transplantation (HCT) for patients 18 years and older, randomized between haplo-cord search and matched unrelated donor (MUD) search for patients with acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS)

DETAILED DESCRIPTION:
Primary Objectives

To compare time from formal search to hematopoietic cell transplantation (HCT) for patients 18 years and older, randomized between haplo-cord search and matched unrelated donor (MUD) search for patients with acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS)

Secondary Objectives

* To compare the percentage of patients who undergo HCT in each study cohort
* To evaluate overall survival from time to randomization by study cohort

ELIGIBILITY:
Inclusion Criteria for Search Phase:

1. Diagnosis of acute myeloid leukemia (AML) or high or very high-risk MDS by international prognostic scoring system revised for whom transplant is recommended
2. 18 years of age or older
3. Subject is likely to be considered for allogeneic transplant in the opinion of the transplant physician (based on age of patient, health, cytogenetics, and/or molecular characteristics).
4. Karnofsky Performance Status (KPS) >/= 70% at time of enrollment. An exception will be made for those with lower KPS at enrollment with an acute worsening that is likely to resolve in the treating physicians judgment (e.g., reversible infection,trauma, medication reaction, etc)
5. Ability to understand and the willingness to sign a written informed consent document for the Search Phase.
6. Patient willing to consider HCT
7. A preliminary search has identified:

   1. An appropriate minimum 4/6 matched umbilical cord unit at intermediate resolution at HLA-A and B, and high resolution at HLA-DRB with a cell dose above 1 x 10(7) TNC/kg for a single umbilical cord blood (UCB) transplant AND
   2. At least one potential 8/8 HLA-matched (HLA-A, -B, -C, and -DRB1) unrelated donor with a probability of 70% AND
   3. Availability of a potential related haploidentical donor.

Exclusion Criteria for Search Phase:

1. Prior formal search was instituted
2. Diagnosis of acute promyelocytic leukemia (APL)
3. Known HLA matched related donor without contraindications to donate
4. Life expectancy severely limited by concomitant illness or uncontrolled infection

Inclusion Criteria for Transplant Phase

1. High-risk AML for which transplant is recommend based on cytogenetic, molecular and morphologic features. Patients must meet institutional standards for disease control prior to transplant.
2. For MDS. IPSS-revised criteria of high or very high at diagnosis.
3. Subject meets institutional criteria for transplant and has acceptable organ and marrow function as defined below:

   1. Serum bilirubin < 2.0mg/dL unless Gilberts disease
   2. Creatinine Clearance > 45 mL/min.1.73m2 as estimated by modified MDRD equation
   3. Left ventricular function 40% or greater
   4. DLCO corrected for hemoglobin >50%
   5. KPS 70% or greater
4. An adequate graft for the defined donor type

   1. Haplo-cord requires a haploidentical adult donor of 14 years of age and at least 50 kg, and a cord blood unit with at least 1.0 x 10(7) TNC/kg and a match of at least 4/6 by intermediate resolution for HLA-A and B and high resolution at DRB1. Donor provides standard of care consent for harvest following institutional policy. Any donor samples or donor research data would be obtained on separate donor research protocol.
   2. For MUD requires a 7/8 or 8/8 HLA matched unrelated donor with high resolution matching at HLA-A, -B, -C, and DRB1. DP matching or DP permissive should be achieved when possible using T-cell epitope strategy.
5. Written informed consent for the transplant phase

Exclusion Criteria for Transplant Phase

1. Life expectancy severely limited by concomitant illness or uncontrolled infection
2. HIV-positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Artz, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Matched Unrelated Donor Search (MUD): If subject meets the inclusion criteria and consents, will undergo a MUD transplant.
  Matched Unrelated Donor Transplant
Period: Overall Study
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD)
Started | 5 | 4
Completed | 2 | 3
Not Completed | 3 | 1
Not completed — No transplant | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD) | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Median (Full Range); unit: years] | 67.9 [53.5 to 71.9] | 61.2 [53 to 66.8] | 62.1 [53 to 71.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Transplant
Description: Time to transplant will be measured from time of date of formal request to stem cell infusion date. Will also capture time from preliminary search to both formal search and transplant date.
Time Frame: Through one year after formal search
Population: We analyze only those who went to transplant.
Measure: Median (Full Range); unit: days
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD)
Number analyzed (Participants) | 2 | 3
days | 69 [63 to 74] | 111 [68 to 149]

2. Secondary Outcome: Percentage of Patients Who Undergo Hematopoietic Cell Transplantation (HCT)
Description: Compare percentage of patients who undergo HCT in each study cohort
Time Frame: Through one year after formal search
Measure: Count of Participants; unit: Participants
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD)
Number analyzed (Participants) | 5 | 4
Participants | 2 | 3

3. Secondary Outcome: Estimated Survival Time
Description: Overall survival time was estimated from date of randomization and from date of transplant using Kaplan-Meier method.
Time Frame: From date of randomization up to 3 years
Population: We analyzed only those who went transplant.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD)
Number analyzed (Participants) | 2 | 3
days
  Days from randomization | 162 [162 to NA] — There are not enough people have died yet to estimate the upper confidence interval. One of two participants survived. | 785 [607 to NA] — There are not enough people have died yet to estimate the upper confidence interval. One of three participants survived.
  Days from transplant | 92 [92 to NA] — There are not enough people have died yet to estimate the upper confidence interval. One of two participants survived. | 673 [467 to NA] — There are not enough people have died yet to estimate the upper confidence interval. One of three participants survived.

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Haplo-Cord Search | Matched Unrelated Donor Search (MUD)
All-Cause Mortality (participants affected / at risk) | 1/2 | 2/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/2 | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Haplo-Cord Search (N=2) | Matched Unrelated Donor Search (MUD) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Weight loss (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-02-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT02648932/Prot_SAP_000.pdf